CLINICAL TRIAL: NCT02721602
Title: Families Preventing Diabetes Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23085
Record Dates: First submitted 2016-02-16; First posted 2016-03-29 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes; Pediatric Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Families in the Families Preventing Diabetes Together intervention group will be asked to participate in four in-person sessions at a local Fairview North metropolitan area clinic over the course of two months. Sessions will focus on age-appropriate nutrition and diabetes education, meal planning and cooking skills, healthful eating, and eating meals as a family. All family members will be asked to attend and will be involved in all four, two-hour sessions. The parent with diabetes will also complete one goal setting telephone call based on motivational interviewing techniques during the intervention period.
  Interventions: Behavioral: Families Preventing Diabetes Together
- Measurement Only (No Intervention): No intervention only measurements

INTERVENTIONS:
Behavioral: Families Preventing Diabetes Together — Families in the intervention group will be asked to participate in four in-person sessions at a local Fairview North metropolitan area clinic over the course of two months. Sessions will focus on age-appropriate nutrition and diabetes education, meal planning and cooking skills, healthful eating, and eating meals as a family. All family members will be asked to attend and will be involved in all four, two-hour sessions. The parent with diabetes will also complete one goal setting telephone call based on motivational interviewing techniques during the intervention period.
  Arms: Intervention Group

SUMMARY:
The current study proposes to study the feasibility and acceptability of the Families Preventing Diabetes Together Intervention among 40 families who have one parent diagnosed with type 2 diabetes and at least 1 child between the ages of 5-14 years of age. Successful recruitment, measurement and randomization of patients and their families will provide data for our aim of assessing feasibility. Patient and family participation in the intervention and feedback via the post-intervention surveys will provide data for our aim of acceptability.

DETAILED DESCRIPTION:
The current study is a randomized controlled trial with 40 families. Twenty families will be randomly assigned to receive usual care consisting of diabetes education delivered through Fairview Health Services. An additional 20 families will be randomized to a family-based, in-person program that focuses on nutrition education, the development of meal planning and cooking skills and promotion of healthful eating for families; the program will augment usual care and diabetes education received from Fairview Health Services for the parent with diabetes. Parents with diabetes who are randomized to the intervention group will also participate in one goal-setting phone call with intervention staff at one point during the intervention program.

Adult patients and their families will be recruited in two ways:

1. from Fairview Health Service's clinics in the North metropolitan area with the assistance of Fairview Health Service diabetes educators, and
2. through MyChart messages informing them about the study.

Adults between the ages of 25 and 55 years who have a diagnosis of Type 2 diabetes, who have participated in at least some diabetes education through Fairview Health Services, and who have at least one child between the ages of 7-12 years of age will be invited to participate in the study. Successful recruitment, measurement and randomization of patients and their families will provide data for our aim of assessing feasibility. Patient and family participation in the intervention and feedback via the post-intervention surveys will provide data for our aim of acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Parent with Type 2 diabetes
* At least 1 child between the ages of 7-12
* Parent has completed at least some Diabetes Education through Fairview Health System

Exclusion Criteria:

* Parent with Type 2 diabetes does not speak or read in English
* No parents with Type 2 diabetes or no children ages 7-12 years
* Parent with Type 2 diabetes has not completed at least some Diabetes Education

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study measured via the ability to successfully recruit 30-40 families for the study. | up to 6 months
  Ability to successfully recruit 30- 40 families in the study will determine feasibility.
Feasibility of the study measured via the ability to successfully measure 100% of the adults and 80% of the children in enrolled families at baseline measurements. | up to 6 months
  Ability to successfully measure 100% of recruited adults and 80% of children in enrolled families at baseline measurements will determine feasibility.
Feasibility of the study measured via the ability to successfully retain 85% of the enrolled families over the course of the study measured by their participate in post-intervention measurements. | up to 6 months
  Feasibility of the study measured via the ability to successfully retain 85% of the enrolled families over the course of the study measured by their participate in post-intervention measurements.
Acceptability of the intervention measured via family participation rates (families attend at least 70% of the sessions). | up to 6 months
  Family participation in the intervention (attending at least 70% of sessions) will determine acceptability.
Acceptability of the intervention measured via family feedback indicating at least 90% approve of the sessions on post-intervention surveys. | up to 6 months
  Acceptability of the intervention measured via family feedback indicating at least 90% approve of the sessions on post-intervention surveys.

SECONDARY OUTCOMES:
Child BMIz | up to 6 months
  Objectively measured height and weight will be used to determine child BMIz values to see if the study resulted in any changes in BMIz between baseline measurements and post-intervention measurements.
Blood glucose control in parent with Type 2 diabetes | up to 6 months
  Change in type 2 diabetic parent's A1C values over the course of the study will be used to measure parent blood glucose control between baseline measurements and post-intervention measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, School of Nursing, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No